CLINICAL TRIAL: NCT05506878
Title: Reduction of Opioid Requirement Associated With Auriculo-Nerve Stimulation Following Open Surgery
Brief Title: Auriculo-Nerve Stimulation on Post-Operative Opioid Requirement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Collaborators: Masimo Corporation (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor of Anesthesiology and Perioperative Medicine and Orthopedic Surgery Director, Regional Anesthesiology Fellowship Program, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY21100077; 1R01DA054513-01A1 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-08-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use; Auriculotherapy; Pain, Abdominal; Cancer Pain; Liver Transplant
Keywords: anesthesiology; auricular neurostimulation; auriculotherapy; open surgery; opioids; pain management
MeSH Terms: conditions — Abdominal Pain; Cancer Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Active device versus Sham Device
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 3 researchers have been appointed to randomization and are not participating in any part of the study other than treatment allocation. The researcher applying the device will not know the treatment allocation, and everyone else (participant, care provider, investigator and outcomes assessor) will be blinded to treatment allocation as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NSS-2 BRIDGE device (Active Comparator): This experimental arm involves the use of the NSS-2 BRIDGE device, which is a disposable device that stimulates the branches of cranial nerves and of the superficial cervical plexus innervating the ear. It will be placed on the subject immediately after surgery and worn for 5 days.
  It is a percutaneous nerve field stimulator (PNFS) system, that can be used as an aid to reduce the symptoms of opioid withdrawal, through application to branches of Cranial Nerves V, VII, IX and X, and the occipital nerves identified by transillumination.
  Interventions: Device: NSS-2 BRIDGE
- Placebo Bridge (Sham Comparator): The sham group involves the use of 3 non-active points, or "nonfunctional points." The sham device will be placed on the subject immediately post-operatively and worn for 5 days just like the active group.
  Interventions: Device: Sham NSS-2 BRIDGE

INTERVENTIONS:
Device: NSS-2 BRIDGE — NBD® will be applied to either the right or left ear in the immediate post-operative setting (PACU). Only a trained and certified research member who has completed the necessary training required by the company will place the device. The individual placing the device will not be involved in any follow up of the subject or any data collection as that researcher will be unblinded to the treatment allocation. The patient, nurses, surgeons, and other members of the research team will all remain blinded to the treatment allocation.
  Once the device is placed, subjects will be asked to perform a "pinch test" throughout the duration of their time wearing the device. To perform the "pinch test" subjects must pinch down on the electrodes and ground to ensure the electrodes are still placed in their designated locations and have not come loose.
  Other Names: Bridge
  Arms: NSS-2 BRIDGE device
Device: Sham NSS-2 BRIDGE — Sham NBD® will be applied to either the left or right ear in the immediate post-operative setting (PACU). Only a trained and certified research member who has completed the necessary training required by the company will place the device. The individual placing the device will not be involved in any follow up of the subject or any data collection as that researcher will be unblinded to the treatment allocation. The patient, nurses, surgeons, and other members of the research team will all remain blinded to the treatment allocation.
  Other Names: Placebo
  Arms: Placebo Bridge

SUMMARY:
The NSS-2 BRIDGE® device (NSS stands for Neuro-Stimulation System) is a disposable device that stimulates the branches of cranial nerves and of the superficial cervical plexus innervating the ear. Because the stimulation of the nerves of the ear by the NSS-2 BRIDGE® device (NBD®) has been shown to modulate pain pathways in rodents, decrease abdominal pain in adolescents with inflammatory bile syndrome and due to the results of our preliminary pilot study, the investigators hypothesized that this technique may also be effective in reducing the requirement for postoperative opioids and provide a non-pharmacological alternative to perioperative opioid use.

To establish the role that the stimulation of the nerves of the ear may have in reducing postoperative opioid requirement, the investigators are proposing to conduct a randomized, placebo controlled study in patients undergoing open abdominal or pelvic surgery requiring at least 5 days of hospitalization. Subjects who have signed an informed consent will be randomized in 2 groups (active NBD® group or inactive NBD® group).

Furthermore, since preoperative and postoperative mood disorders have been shown to increase postoperative pain levels and opioid requirement by up to 50%, the investigators further hypothesize that the stimulation of the ear nerves by the NSS-2 BRIDGE® effects may be in part mediated by a reduction of the level of anxiety, depression and catastrophizing as assessed using validated questionnaires.

DETAILED DESCRIPTION:
It is established that the perioperative prescription of opioids, including doses prescribed after discharge from the hospitals, is an important contributor to the current opioid epidemic. Although many factors have been implicated including history of addiction, mood disorders and the type of surgery, the quantity and duration of opioid treatment play an important role in a patient's development of opioid use disorder (OUD). Despite recommendations by the majority of surgery and anesthesiology professionals to limit the perioperative use of opioids, and to favor the use of non-opioid analgesics, OUD remains a serious concern. Consequently, developing alternative techniques to minimize the perioperative use of opioids is critical in the fight against the current opioid epidemic.

Auriculotherapy, a form of acupuncture is an ancient technique used to treat many conditions, including pain. Its mechanism of action is believed to be primarily via the stimulation of the branches of the vagal, trigeminal, glossopharyngeal, hypogastric, facial and superficial cervical plexus nerves innervating which secondarily modulate the pain pathway and the limbic system at the level of the brainstem, spin and central nervous system. However, the use of auriculotherapy has been limited in part by the requirement for long and specific training and the lack of well-designed clinical trials demonstrating its effectiveness.

This study design is based on the high frequency of OUD following surgery for cancer and the positive results from our exploratory Institutional Review Board (IRB)- approved, randomized and placebo-controlled pilot study that assessed the effects of the NSS-2 BRIDGE® device on perioperative pain and opioid requirement in different surgical oncology models. This was a study that included subjects undergoing both open and laparoscopic procedures of different types of surgeries for abdominal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Scheduled for elective open primary abdominal and pelvic colorectal cancer resection surgical procedures at UPMC Shadyside Hospital, UPMC Magee-Women's Hospital, or UPMC Passavant Hospital and following the standard ERAS protocol. OR scheduled for a living-donor liver transplant surgery at UPMC Montefiore Hospital under the ERAS protocol.
3. Expected hospital stay of approximately 5 days

Exclusion Criteria:

1. Patients who are considered by the medical or surgical team to not be able to give consent
2. Clinical evidence of anxiety, depression, including suicidal ideation. The diagnostic will be based on medical history, the current treatment, and the clinical examination. The PI or Co-I will be the one making the determination to enroll the subject after the subject undergoes psychosocial testing included in the protocol and that corresponding scores have been established. These tests will only be conducted after the patient has signed an informed consent form.
3. Chronic pain condition that at the discretion of the PI, should exclude the subject from participating -or- chronic opioid use defined as daily use of 60 mg of oral opioid equivalent. The diagnostic will be based on the medical history, the current treatment, and the clinical examination. The PI or Co-I will be the one making the determination to enroll the subject.
4. True allergy to all opioid medications. The diagnostic will be based on the medical history, and the determination of the symptoms associated with the recorded allergy. The PI or Co-I will be the one making the determination to enroll the subject.
5. History of or current alcohol abuse (defined as daily use of more than 1 liter of wine and/or 3 or more shots of hard liquor) or drug abuse (defined as daily use of illicit drugs) for at least 3 months. The PI or Co-I will be the one making the determination to enroll the subject.
6. Surgical procedure performed laparoscopically
7. Non elective surgery
8. Pregnancy
9. Contraindication for use of NBD® (including patients with cardiac pacemaker, hemophilia, and psoriasis vulgaris diagnosis and/or ear eczema)
10. Patients intubated with sedation, and/or receiving fentanyl infusion for sedation post-surgery.
11. Rapid recovery surgeries
12. Subjects with a diagnosed seizure disorder
13. Use of dexmedetomidine in the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | (OME) at 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-operative
  Assess how the use of the NSS-2 BRIDGE Device over 5 days stimulation period affect the participant's total opioid consumption using morphine equivalent following an open abdominal or pelvic surgery.

SECONDARY OUTCOMES:
Post-operative pain rating using a numerical rating scale | 1 hour post NBD placement, days 1,2,3,4,5 post-operative, 1 month post-operative, 3 months post-operative
  Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome.
Area under the curve of post-operative pain rating using a numerical rating scale | 1 hour post NBD placement, days 1,2,3,4,5 post-operative, 1 month post-operative, 3 months post-operative
  Area under the curve of Numerical Rating Scale (NRS) Pain scores on a scale from 0-10, with 0 being no pain, 5 being moderate pain and 10 being the worst imaginable pain. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome, between 1-hour post NBD placement and day 5
Post-operative nausea and vomiting rating | 1 hour post NBD placement, days 1, 2, 3, 4, & 5 post-operative
  Numerical Rating Scale (NRS) nausea scores on a scale from 0-10, with 0 being no nausea, 5 being moderate nausea and 10 being the worst imaginable nausea and vomiting. The lowest possible score is 0 and the highest possible score is 10. Higher scores represent a worse outcome.
Pre-operative emotional distress related to anxiety | Baseline, pre-surgery
  Pre-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the Patient Reported Outcome Measurement Information System (PROMIS) Emotional Distress -Anxiety- Short Form 8a questionnaire prior to surgery. There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative change in emotional distress related to anxiety | Day 1, 2, 3, 4, 5, 1 month, and 3 months post-operative
  Post-operative emotional distress related to anxiety will be measured by assessment of participant's answers to the PROMIS Emotional Distress -Anxiety- Short Form 8a questionnaire.There are 8 questions about how the participants may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative emotional distress related to depression | Baseline, pre-surgery
  Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Post-operative change in emotional distress related to depression | Day 1, 2, 3, 4, 5, 1 month, and 3 months post-operative
  Pre-operative emotional distress related to depression will be measured by assessment of participant's answers to the PROMIS Emotional Distress-Depression-Short Form questionnaire prior to surgery. There are 8 questions about how the participant may have felt in the past 7 days. The scale for each question is from 1, never felt this way in the past 7 days, to 5, always have felt this way in the past 7 days. The overall questionnaire scores can range from 8 (least severe score) to 40 (most severe score). Higher scores present a worse outcome.
Pre-operative sleep disturbance | Baseline, pre-surgery
  Pre-operative sleep disturbance will be measured by assessment of the participant's answers to the PROMIS item Bank v1.0 - Sleep Disturbance - Short Form 8a. There are 8 questions about how the participant may have felt about their sleep quality in the past 7 days. The scale for 1 question is very poor in the past 7 days to very good in the past 7 days. The scale for 7 questions is not at all in the past 7 days to very much in the past 7 days.
Post-operative change in sleep disturbance | Day 1, 2, 3, 4, 5, 1 month, and 3 months post-operative
  Post-operative sleep disturbance will be measured by assessment of the participant's answers to the PROMIS item Bank v1.0 - Sleep Disturbance - Short Form 8a. There are 8 questions about how the participant may have felt about their sleep quality in the past 7 days. The scale for 1 question is very poor in the past 7 days to very good in the past 7 days. The scale for 7 questions is not at all in the past 7 days to very much in the past 7 days.
Pre-operative pain rating using the Pain Catastrophizing Scale | Baseline, pre-surgery
  Pre-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome
Change in post-operative pain rating using the Pain Catastrophizing Scale | Day 1, 2, 3, 4, 5, 1 month, and 3 months post-operative
  Post-operative pain ratings will be measured by the assessment of the participant's answers to the Pain Catastrophizing Scale questionnaire. There are 14 statements related to pain that participants will record experiencing on a scale of 0 being experienced not at all to 4 being experienced all of the time. The lowest possible score is 0 and the highest possible score is 56. Higher scores present a worse outcome
Pre-operative Brief Symptom Index Somatization Scale | Baseline, pre-surgery
  The Brief Symptom Index Somatization Scale measures the participant's distress about 6 symptoms. There are 6 symptoms that the participant rates according to their level of stress. The symptoms include: faintness or dizziness, pains in heart or chest, nausea or upset stomach, trouble getting your breath, numbness or tingling, and feeling weak. The subject may select one of 5 responses: not at all, a little bit, moderately, quite a bit, and extremely.
Change in the Brief Symptom Index Somatization Scale | Day 1, 2, 3, 4, 5, 1 month, and 3 months post-operative
  The Brief Symptom Index Somatization Scale measures the participant's distress about 6 symptoms. There are 6 symptoms that the participant rates according to their level of stress. The symptoms include: faintness or dizziness, pains in heart or chest, nausea or upset stomach, trouble getting your breath, numbness or tingling, and feeling weak. The subject may select one of 5 responses: not at all, a little bit, moderately, quite a bit, and extremely.
Time to Oral Intake | Day of surgery up to 5 days
  Evaluate time to oral intake post-operative.
Time to Ambulation | Day of surgery up to 5 days
  Evaluate time to ambulation, walking greater than 15 feet
Time to discharge from the recovery unit | Day of surgery up to 5 days
  Evaluate the time to discharge from the recovery unit (PACU) post-operatively
Length of hospital stay | Day of surgery up to 30 days
  Evaluate time to hospital discharge from out of OR time
Device tolerability | Time of device placement, 1 hour after placement, 6, 12, 18, 24, 48, 72, 96, and 120 hours post-operative
  Participants will rate on a scale of 0 to 10, 0 being completely tolerable and 10 being completely intolerable.
Overall Patient Satisfaction | Day of Surgery through discharge or post-operative day 30, whichever comes first
  Participants will be asked to assess their overall satisfaction upon discharge on a scale of 0 (least satisfaction) to 10 (highest satisfaction) at the time of discharge
Total Opioid Consumption | Post-operative day 5, 1-month, and 3-months post-operative
  Participant opioid consumption will be recorded using an e-Pill time cap dispenser which records the date and time at which opioids were taken.
Prescription Drug Monitoring Program (PDMP) | Post-operative day 30
  Participant PDMP will be reviewed to determine the average number of opioid refill requests by the subjects.
Prescription Drug Monitoring Program (PDMP) | Post-operative day 60
  Participant PDMP will be reviewed to determine the average number of opioid refill requests by the subjects.
Prescription Drug Monitoring Program (PDMP) | Post-operative day 90
  Participant PDMP will be reviewed to determine the average number of opioid refill requests by the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, PhD, MBA, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - University of Pittsburgh Medical Center - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Passavant Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
There will be annual NIH reports, and publicly sharing de-identified data with NIH.
Supporting Information: CSR
Time Frame: Every 6 months for 4 years.
Access Criteria: The PI will be ultimately responsible for coordinating, obtaining and sharing de-identified Electronic Health Record (EHR)-based and electronically reported and prospectively collected clinical and outcome data.